CLINICAL TRIAL: NCT06221982
Title: Transjugular Intrahepatic Portosystemic Shunt for Patients With Portal Hypertension: an Observational, Cohort Study
Brief Title: TIPS for PH Patients: an Observational, Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-005
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Cirrhosis Portal
Keywords: Transjugular intrahepatic porsystemic shunt
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing TIPS procedure: Patients undergoing TIPS procedure due to portal hypertension-related complications
  Interventions: Other: No intervention, observational study

INTERVENTIONS:
Other: No intervention, observational study — Observational study, no intervention

SUMMARY:
This is a single-center, prospective, observational study intended to include patients receiving TIPS for portal hypertension. Baseline data of enrolled patients were recorded, and samples of ascites, feces and urine were collected before surgery. Venous blood (superior mesenteric vein, hepatic vein, peripheral vein) from different parts of the entero-hepatic axis was retained during operation, and patients were followed up regularly for 2 years. The incidence of infection, hepatic encephalopathy, upper gastrointestinal hemorrhage and ascites in patients with portal hypertension who received TIPS intervention were observed within 3 months after operation. And the stent patency was observed within 2 years after surgery. To investigate the characteristics of microbial, protein and metabolic components on enterohepatic axis and their relationship with prognosis of patients with cirrhosis by detecting microbiome, proteome and metabolome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing TIPS due to complications related to portal hypertension；
2. Age between 18 to 85 years;
3. Signed informed consent;

Exclusion Criteria:

1. Combined with liver cancer (out of the Milan criteria) or combined with other organ malignancies which had less than 3 months of expected survival;
2. Combined with severe cardiopulmonary disease (severe pulmonary hypertension and heart failure or severe heart valve insufficiency or renal insufficiency), the expected survival is less than 3 months;
3. Failure of TIPS procedure;
4. Women who plan to become pregnant or who are pregnant or breastfeeding；
5. Conditions deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing TIPS due to complications related to portal hypertension；
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
TIPS shunt dysfunction | two years

SECONDARY OUTCOMES:
death | 2 years
liver transplant | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang hospital, Southern Medical Uiversity, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No